CLINICAL TRIAL: NCT02898662
Title: A Phase 2 Placebo-Controlled, Randomized, Double Blind, Adaptive Dose Trial of the Safety and Efficacy of Inhaled AZD1419 in Adults With Eosinophilic, Moderate to Severe Asthma
Brief Title: AZD1419 Ph2a Study
Acronym: INCONTRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2500C00003
Record Dates: First submitted 2016-08-16; First posted 2016-09-13 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Asthma
Keywords: inhaled; TLR9 agonist; withdrawal design; loss of control
MeSH Terms: conditions — Asthma; Respiratory Aspiration | interventions — AZD1419

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD1419 (Experimental): Dose adaption of AZD1419, 4 mg or 8 mg or 1 mg based on occurence of AE's
  Interventions: Drug: AZD1419
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1419 — Inhaled AZD1419 administered at the clinic as once weekly inhalations with the I-neb® device. Start dose is 4 mg and dose adaptation is applied (downtitration to 1mg or uptitration to 8 mg or remain on 4 mg) based on appearance of flu like adverse events
  Arms: AZD1419
Drug: Placebo — Inhaled Placebo administered at the clinic as once weekly inhalations with the I-neb® device. Start dose is Placebo 4 mg and dose adaptation is applied (downtitration to 1mg or uptitration to 8 mg or remain on 4 mg) based on appearance of flu like adverse events
  Arms: Placebo

SUMMARY:
Ph2a study planned to be run at approximately 16-18 sites in 4 EU countries (Denmark, Hungary, Poland and Sweden) enrolling approximately 170 patients to ensure 70 randomized patients with eosinophilic, moderate to severe asthma. The patients will receive 13 once weekly inhaled doses of the study drug. Treatment is initiated on top of their ICS/LABA controller medication, which is then tapered down and withdrawn during a period of 3 weeks and during the last 3 weeks of treatment the study drug is given as monotherapy. SABA is used as reliever medication during the whole study period. Primary endpoint is Loss of asthma control. When the endpoint is met, patients will resume their ICS/LABA, will be followed for an additional 4 weeks and will thereafter discontinue the study.

DETAILED DESCRIPTION:
Ph2a study planned to be run in approximately 16-18 sites in 4 EU countries (Denmark, Hungary, Poland and Sweden) enrolling approximately 170 patients to ensure 70 randomized patients with eosinophilic, moderate to severe asthma.

The study has a withdrawal design.The patients will receive 13 once weekly inhaled doses of the study drug (AZD1419 or placebo). Treatment is initiated with 6 doses of the study drug on top of their ICS/LABA controller medication. Prior to the 7th dose of the study drug the LABA is withdrawn. The following 3 doses are given when ICS is tapered down. Dose 7 is given on top of 100% of their ICS, dose 8 is given on top of 50% of the ICS dose, which is then tapered down to 25% the following week and withdrawn completely prior to dose 10 of the study drug. During the last 3 weeks of treatment (ie last 4 doses), the study drug is given as monotherapy. SABA is used as reliever medication during the whole study period. Primary endpoint is Loss of asthma control, defined as any of the following criteria: a) An increase of ACQ-5 to 1.5 or more b) A reduction of 30% or more in morning peak expiratory flow (PEF) from baseline on 2 consecutive days c) At least six additional reliever inhalations of SABA in a 24-hour period relative to baseline on 2 consecutive days and d) An exacerbation requiring systemic corticosteroids

When the endpoint is met, patients will resume their regular ICS/LABA controller medication and will be followed for an additional 4 weeks, when they do an Early Discontinuation (ED) Visit and will thereafter leave the study. For patients not loosing their asthma control, the full Observational period is up to week 52, when they will do an End of Treatment Visit (EOT). Study procedures are the same on ED and EOT Visits.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years and above
* Physician-diagnosed asthma requiring treatment with ICS and a long-acting beta agonist (LABA). Patients must have taken ICS plus LABA controller medication for at least 3 months prior to screening
* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) ≥50% predicted
* Female patients must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception
* Male patients must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) from the first dose of the IMP and until 1 month after the last dose of the IMP to prevent pregnancy in a partner
* Blood eosinophil levels ≥ 250 cells/μL at screening OR a history of blood eosinophil levels ≥ 250 cells/μL at any time in the preceding 2 years AND blood eosinophil levels ≥ 150 cells /μL at screening. The eosinophilia must be believed to be due to asthma and not have other known causes, e.g. helminth infection
* ACQ-5 score ≤1.5 at screening
* ACQ-5 score ≤0.75 at randomization
* Documentation of any of the following within 5 years prior to Visit 1:

  * Proof of post-bronchodilator reversibility in FEV1 of ≥12% and ≥200 mL
  * Proof of a positive response to a methacholine or histamine challenge (a decrease in FEV1 by 20% [PC20] at ≤8 mg/mL)
  * Proof of positive response to mannitol challenge (a decrease in FEV1 by 15% [PD15] at ≤635 mg or a >10% decrease in FEV1 between consecutive doses)
  * Proof of diurnal variability in PEF >20% over the course of 24 hours in at least 4 out of 7 consecutive days If historical documentation is not available, proof of reversibility or a positive response to a methacholine, histamine or mannitol challenge or diurnal variation must be demonstrated according to above and documented during Visit 1

Exclusion Criteria:

* Clinically significant lung disease other than asthma (eg, chronic obstructive pulmonary disease, cystic fibrosis, allergic bronchopulmonary aspergillosis, active tuberculosis).
* History of autoimmune disease including but not limited to Wegener's granulomatosis, system lupus erythematosus, rheumatoid arthritis, Sjögren's syndrome, multiple sclerosis, autoimmune thrombocytopenia, primary biliary cirrhosis or any other autoimmune disease considered clinically relevant by the investigator
* Ongoing allergen immunotherapy or plans to begin such therapy during the study period
* DLco ≤ 60% of the lower limit of normal
* Breast feeding, pregnancy or intention to become pregnant during the course of the study
* Changes in chest X-ray suggesting clinically significant parenchymal disease other than asthma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Denmark (4):
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Næstved
  - Research Site, Odense C
- Hungary (5):
  - Research Site, Balassagyarmat
  - Research Site, Edelény
  - Research Site, Farkasgyepü
  - Research Site, Miskolc
  - Research Site, Törökbálint
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Lubin
- Sweden (3):
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Stockholm

REFERENCES:
- See also: Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2500C00003&attachmentIdentifier=d303e80b-f6fb-4d86-8aaa-b300ca034443&fileName=Final-D2500C00003-csp-v3.pdf&versionIdentifier=
- See also: Statistical Analysis Plan (SAP) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D2500C00003&attachmentIdentifier=819b73ac-d738-44a9-82c9-1fe901aaec61&fileName=d2500c00003-sap-ed-2.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 16 centers in 4 countries (Hungary, Poland, Denmark and Sweden) between 12 October 2016 and 25 September 2018. Participants with eosinophilic moderate to severe asthma on a maintenance treatment of controller inhaled corticosteroids (ICS) + long-acting β2 agonists (LABA) and no other controller medication were recruited.
Pre-assignment Details: The study had a screening period (2-4 weeks), a 12-week dosing period and an observation period (up to 40 weeks). A total of 81 participants were randomized in this study to test the hypothesis that AZD1419 provided sustained asthma control in eosinophilic asthma participants after removal of ICS and LABA medication.
Groups:
- AZD1419: Participants received AZD1419 for inhalation via nebuliser solution (up to 13 doses). All participants received 4 milligrams (mg) AZD1419 once weekly for 4 doses. The following 9 doses were adapted based on tolerability (severity of flu-like symptoms). Participants were prescribed their usual controller medication (ICS + LABA) in separate inhalers. During the dosing period, controller medications were gradually reduced and discontinued. Treatment was initiated with 6 doses of AZD1419 on top of the participant's controller medication, LABA was then stopped on the evening prior to receiving dose 7, and ICS was gradually tapered down and discontinued during the next 3 weeks before being discontinued in the evening prior to receiving AZD1419 dose 10.
- Placebo: Participants received placebo for inhalation via nebuliser solution (up to 13 doses). All participants received placebo to match 4 mg AZD1419 once weekly for 4 doses. The following 9 doses were adapted based on tolerability (severity of flu-like symptoms). Participants were prescribed their usual controller medication (ICS + LABA) in separate inhalers. During the dosing period, controller medications were gradually reduced and discontinued. Treatment was initiated with 6 doses of placebo on top of the participant's controller medication, LABA was then stopped on the evening prior to receiving dose 7, and ICS was gradually tapered down and discontinued during the next 3 weeks before being discontinued in the evening prior to receiving placebo dose 10.
Period: Overall Study
Arm/Group | AZD1419 | Placebo
Started | 40 | 41
Completed Treatment | 25 | 29
Completed (Completed the study) | 11 | 13
Not Completed | 29 | 28
Not completed — Adverse Event | 1 | 0
Not completed — Loss of asthma control | 23 | 24
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Technical issue | 0 | 1
Not completed — Randomized in error | 0 | 1
Not completed — Subject decision | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received any investigational product (IP), irrespective of their protocol adherence and continued participation in the study.
Groups:
- AZD1419: Participants received AZD1419 for inhalation via nebuliser solution (up to 13 doses). All participants received 4 mg AZD1419 once weekly for 4 doses. The following 9 doses were adapted based on tolerability (severity of flu-like symptoms). Participants were prescribed their usual controller medication (ICS + LABA) in separate inhalers. During the dosing period, controller medications were gradually reduced and discontinued. Treatment was initiated with 6 doses of AZD1419 on top of the participant's controller medication, LABA was then stopped on the evening prior to receiving dose 7, and ICS was gradually tapered down and discontinued during the next 3 weeks before being discontinued in the evening prior to receiving AZD1419 dose 10.
- Total: Total of all reporting groups
Arm/Group | AZD1419 | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (13.3) | 53.3 (15.4) | 55.3 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 40 | 40 | 80
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Events for Time to Loss of Asthma Control (LOAC) up to Week 52 - Cox Regression Analysis
Description: LOAC was defined as any of the following:
  * Increase of asthma control questionnaire-5 (ACQ-5) to ≥ 1.5.
  * ≥ 30% reduction in morning peak expiratory flow (PEF) from baseline on 2 consecutive days.
  * ≥ 6 additional reliever inhalations of short-acting β agonist (SABA) in a 24-hour period relative to baseline on 2 consecutive days.
  * Exacerbation requiring systemic corticosteroids as decided by Investigator. Time to LOAC was calculated as start date of first LOAC - date of randomization + 1. Start date of LOAC was latest date that 1 of the 4 criteria were satisfied immediately prior to the exacerbation start date, provided no more than 7 days between LOAC and exacerbation start date. Time to LOAC was displayed using a Kaplan-Meier plot and the outcome measure is presented as number of participants with events. Cox regression analysis was used to compare treatments.
Time Frame: Baseline (Week 0) up to Week 52
Population: The FAS included all randomized participants who received any IP, irrespective of their protocol adherence and continued participation in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 40 | 41
Participants | 24 | 24
Statistical Analysis 1: Comparison: AZD1419 vs Placebo; Comparison between groups for time to LOAC. Cox regression model analysis with age and gender included as covariates; Test type: Other — The null hypothesis was that during the 52-week double-blind treatment period, the time to LOAC in the AZD1419 arm was equal to the corresponding time to LOAC in the placebo arm; p = 0.5722, Regression, Cox — 1-sided p-value; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.59 to 1.87] — Hazard ratio < 1 favours AZD1419 over placebo

2. Secondary Outcome: Number of Participants Experiencing LOAC up to Week 52 - Generalized Estimating Equation Analysis
Description: LOAC was defined as any of the following:
  * Increase of ACQ-5 to ≥ 1.5.
  * ≥ 30% reduction in morning PEF from baseline on 2 consecutive days.
  * ≥ 6 additional reliever inhalations of SABA in a 24-hour period relative to baseline on 2 consecutive days.
  * Exacerbation requiring systemic corticosteroids. Number of participants experiencing LOAC up to Week 52 is presented. A generalized linear model based on a generalized estimating equation was used to compare treatments.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 40 | 41
Participants | 24 | 24
Statistical Analysis 1: Comparison: AZD1419 vs Placebo; Comparison between groups for participants experiencing LOAC. Odds ratio was estimated using a generalized linear model based on a generalized estimating equation approach fitting treatment, visit and age and gender as covariates; Test type: Other; p = 0.2006, Generalized estimating equation analysis — 2-sided p-value; Odds Ratio (OR) = 1.86, 95% CI 2-sided [0.72 to 4.79]

3. Secondary Outcome: Least Squares (LS) Mean ACQ-5 Score Over 52 Weeks
Description: In the ACQ-5 questionnaire, participants were asked to recall the status of their asthma during the previous week with regards to symptoms. The questionnaire included the items:
  * Awoken at night by asthma symptoms.
  * Severity of asthma symptoms in the morning.
  * Limitation of daily activities due to asthma.
  * Shortness of breath.
  * Wheeze. The ACQ-5 score was computed as the un-weighted mean of responses to the 5 items, measured on a 7-point scale from 0 (totally controlled) to 6 (severely uncontrolled). A lower score indicated a better outcome. If ACQ-5 reached a value of 1.5 or more, the participant was reported as having LOAC. Estimates of the LS mean over 52 weeks were analyzed using a repeated measures analysis with treatment, baseline ACQ-5, week and treatment-by-week with participant as random effects, and age and gender as covariates. Baseline was the average of non-missing daily measures/scores over the last 5 days prior to and including the morning of randomization.
Time Frame: Baseline (Week 0) up to Week 52
Population: The FAS included all randomized participants who received any IP, irrespective of their protocol adherence and continued participation in the study. Only participants with data available for analysis are presented.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 37 | 41
scores on a scale | 0.56 (0.07) | 0.59 (0.07)
Statistical Analysis 1: Comparison: AZD1419 vs Placebo; Comparison between groups for ACQ-5 score. Repeated measures analysis; Test type: Other; p = 0.8166, Repeated measures analysis — 2-sided p-value; LS Mean difference = -0.02, 95% CI 2-sided [-0.22 to 0.17]

4. Secondary Outcome: LS Mean Asthma Daily Diary Score (Weekly Total) Over 52 Weeks
Description: Asthma symptoms during night-time and daytime were recorded by the participant each morning and evening in the Asthma Daily Diary. Symptoms were recorded using a 4-point response scale, which ranged from 0 to 3, where 0 indicated no asthma symptoms. Asthma symptom daytime score (recorded in the evening), night-time score (recorded in the morning), and total score were calculated separately. The daily asthma symptom total score was calculated by taking the sum of the night-time and daytime asthma symptom scores recorded each day, ranging from 0 to 6. A lower symptom score indicated a better outcome. Estimates of the LS mean over 52 weeks were analyzed using a repeated measures analysis with treatment, baseline asthma daily diary weekly average, week and treatment-by-week with participant as random effects, and age and gender as covariates. Baseline was the average of non-missing daily measures/scores over the last 5 days prior to and including the morning of randomization.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 38 | 41
scores on a scale | 0.79 (0.10) | 0.82 (0.10)
Statistical Analysis 1: Comparison: AZD1419 vs Placebo; Comparison between groups for asthma daily diary score. Repeated measures analysis; Test type: Other; p = 0.8412, Repeated measures analysis — 2-sided p-value; LS Mean difference = -0.03, 95% CI 2-sided [-0.32 to 0.26]

5. Secondary Outcome: Number of Participants With Events for Time to Moderate Or Severe Exacerbation up to Week 52
Description: Moderate exacerbation was defined as a temporary increase in maintenance therapy to prevent a severe event supported by sustained (≥ 2 day) worsening in at least 1 key control metric ie, asthma score, reliever medication use, night time awakening or morning PEF.
  Severe exacerbation was defined as a worsening in asthma symptoms and:
  * Use of systemic corticosteroids for at least 3 days and/or
  * An unscheduled or emergency room visit due to asthma symptoms requiring systemic corticosteroids and/or
  * An in-patient hospitalization due to asthma requiring systemic corticosteroids. Time to moderate or severe asthma exacerbation was calculated as start date of first moderate or severe exacerbation - date of randomization + 1. Time to moderate or severe asthma exacerbation was displayed using a Kaplan-Meier plot and the outcome measure is presented as number of participants with events.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 40 | 41
Participants | 13 | 16
Statistical Analysis 1: Comparison: AZD1419 vs Placebo; Comparison between groups for time to moderate or severe asthma exacerbation. Cox regression model analysis with age and gender included as covariates; Test type: Other — The null hypothesis was that the time to moderate or severe exacerbation was not different between AZD1419 and placebo; p = 0.5477, Regression, Cox — 2-sided p-value; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.38 to 1.67] — Hazard ratio < 1 favours AZD1419 over placebo
Statistical Analysis 2: Comparison: AZD1419 vs Placebo; Comparison between groups for participants with moderate or severe asthma exacerbation. Odds ratio was estimated using a generalized linear model based on a generalized estimating equation approach fitting treatment and visit as covariates; Test type: Other; p = 0.7294, Generalized estimating equation analysis — 2-sided p-value; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.41 to 1.86]

6. Secondary Outcome: Percentage of Participants Using Reliever Medication up to Week 52
Description: The use of SABAs was allowed as rescue medication (reliever bronchodilator) throughout the study. Reliever medication use was captured in the Asthma Daily Diary twice daily (morning and evening), recorded as the number of inhaler puffs. The number of inhalations (puffs) per day was calculated as: number of night inhaler puffs + number of day inhaler puffs. Percentage of participants using reliever medication (SABA) up to Week 52 is presented.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 40 | 41
percentage of participants | 100 | 100

7. Secondary Outcome: LS Mean Pre- and Post-Bronchodilator (BD) Forced Expiratory Volume in 1 Second (FEV1) Over 52 Weeks
Description: Lung function was assessed by pre- and post-BD FEV1 which was measured by spirometry. To ensure quality control, all spirometry measurements were reviewed to ensure that they met American Thoracic Society / European Respiratory Society criteria for acceptability. Estimates of the LS mean over 52 weeks were analyzed using a repeated measures analysis with treatment, baseline FEV1 (pre- or post-BD, as applicable), visit and treatment-by-visit with participant as random effects, and age and gender as covariates. Baseline was the last non-missing measurement recorded prior to randomization.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 37 | 39
Liters
  pre-BD FEV1 | 2.24 (0.05) | 2.18 (0.05)
  post-BD FEV1 | 2.36 (0.05) | 2.39 (0.05)
Statistical Analysis 1: Comparison: AZD1419 vs Placebo; Comparison between groups for pre-BD FEV1. Repeated measures analysis; Test type: Other; p = 0.3764, Repeated measures analysis — 2-sided p-value; LS Mean difference = 0.06, 95% CI 2-sided [-0.08 to 0.20]
Statistical Analysis 2: Comparison: AZD1419 vs Placebo; Comparison between groups for post-BD FEV1. Repeated measures analysis; Test type: Other; p = 0.7013, Repeated measures analysis — 2-sided p-value; LS Mean difference = -0.03, 95% CI 2-sided [-0.17 to 0.11]

8. Secondary Outcome: LS Mean Total PEF (Weekly) Over 52 Weeks
Description: Morning and evening PEF measurements were recorded by the participant on a daily basis and then averaged over the week. The weekly average total PEF was calculated by taking the sum of the average of the weekly morning mean and weekly evening mean. Estimates of the LS mean over 52 weeks were analyzed using a repeated measures analysis with treatment, baseline PEF, week and treatment-by-week with participant as random effects, and age and gender as covariates. Baseline was the average of non-missing daily measures/scores over the last 5 days prior to and including the morning of randomization.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Liters/minute
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 38 | 41
Liters/minute | 325.33 (5.77) | 325.65 (5.79)
Statistical Analysis 1: Comparison: AZD1419 vs Placebo; Comparison between groups for PEF. Repeated measures analysis; Test type: Other; p = 0.9686, Repeated measures analysis — 2-sided p-value; LS Mean difference = -0.32, 95% CI 2-sided [-16.54 to 15.90]

9. Secondary Outcome: LS Mean Fractional Exhaled Nitric Oxide (FeNO) (Weekly) Over 52 Weeks
Description: FeNO measurements were taken at home by participants every second day. The weekly average FeNO was based on the average of measurements taken at home for a specific week. Estimates of the LS mean over 52 weeks were analyzed using a repeated measures analysis with treatment, baseline FeNO, week and treatment-by-week with participant as random effects, and age and gender as covariates. Baseline was the average of non-missing daily measures/scores over the last 5 days prior to and including the morning of randomization.
Time Frame: Baseline (Week 0) up to Week 52
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: parts per billion
Arm/Group | AZD1419 | Placebo
Number analyzed (Participants) | 35 | 38
parts per billion | 33.26 (2.33) | 35.28 (2.33)
Statistical Analysis 1: Comparison: AZD1419 vs Placebo; Comparison between groups for FeNO. Repeated measures analysis; Test type: Other; p = 0.5403, Repeated measures analysis — 2-sided p-value; LS Mean difference = -2.02, 95% CI 2-sided [-8.55 to 4.52]

ADVERSE EVENTS:
Time Frame: From first dose of IP (Week 0) up to Week 52.
Description: The safety analysis set included all participants who received any IP.
Arm/Group | AZD1419 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 3/40 | 1/41
Other Adverse Events (participants affected / at risk) | 22/40 | 11/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1419 (N=40) | Placebo (N=41)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary eosinophilia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD1419 (N=40) | Placebo (N=41)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Chills (General disorders) | 6 (13) | 1 (1)
Pyrexia (General disorders) | 10 (22) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (13) | 1 (2)
Headache (Nervous system disorders) | 6 (9) | 4 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT02898662/SAP_001.pdf
  • Study Protocol (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT02898662/Prot_002.pdf